CLINICAL TRIAL: NCT05698316
Title: A Collaborative Resource of Heidelberg Multimodal Imaging of Intermediate and Early Atrophic AMD Cases to Study Prediction of Disease Progression: (INTERCEPT-AMD)
Brief Title: A Collaborative Resource of Heidelberg Multimodal Imaging of Intermediate and Early Atrophic AMD Cases to Study Prediction of Disease Progression
Acronym: INTERCEPT-AMD
Status: Active, not recruiting | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: ECR-AMD-2023-14
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Age Related Macular Degeneration; Intermediate AMD; Atrophy; Prediction
MeSH Terms: conditions — Macular Degeneration; Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age related macular degeneration: Collection of both retrospective and prospective data collection in 3 visits.
  Interventions: Diagnostic Test: Collection of both retrospective and prospective data collection in 3 visits.

INTERVENTIONS:
Diagnostic Test: Collection of both retrospective and prospective data collection in 3 visits. — 3 clinic visits with multimodal imaging done at least at 6 months interval between 2 visits and meet the inclusion and exclusion criteria. Those with one visit remaining to complete 2 years, images will be acquired prospectively. In addition to the images, routine demographic data (age and sex) and available visual acuity (VA) (BCVA if possible, VA with Pinhole or VA with patient's glasses) will be collected. Multimodal imaging includes mandated macular OCT with or without enhanced depth imaging and infrared imaging. Fundus autofluorescence (AF) and multicolor imaging are optional. All imaging must be done on Heidelberg Spectralis system.

SUMMARY:
This is a multicentre retrospective and prospective cohort study with the goal to develop a well-characterised multimodal image database of eyes with intermediate AMD with and without early atrophy. The main objectives are:

1. Develop a collaborative well-characterised database on intermediate AMD with or without early atrophy.
2. Grading of these images to explore imaging markers of progression.
3. Develop predictive models as a secondary analysis of our dataset.

This study will recruit around 1.000 eyes in 6 months. All consenting patients who have had at least 3 clinic visits with multimodal imaging done at least at 6 months interval between 2 visits and meet the inclusion and exclusion criteria will be included in the study for retrospective data collection. Those with one visit remaining to complete 2 years, images will be acquired prospectively. In addition to the images, routine demographic data (age and sex) and available visual acuity (VA) (BCVA if possible, VA with Pinhole or VA with patient's glasses) will be collected. Multimodal imaging includes mandated macular OCT with or without enhanced depth imaging and infrared imaging. Fundus autofluorescence (AF) and multicolor imaging are optional. All imaging must be done on Heidelberg Spectralis system.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the commonest cause of visual impairment in older people in Europe. It is a slowly progressing complex disorder. The clinical progression is best described as early, intermediate, and advanced based on the latest classification system on colour fundus photographs. However, multimodal imaging has enabled visualisation of further changes in the retina on optical coherence tomography (OCT), infrared imaging, and autofluorescence. So, a large database of imaging data of intermediate AMD will facilitate researchers to study the disease progression in detail. This study is a collaborative effort by investigators across many Member Sites in Europe that are members of EVICR.net to pool datasets for secondary analysis.

EVICR.net is a network of Ophthalmological Clinical Research Sites, dedicated to performing multinational clinical research in ophthalmology with the highest standards of quality, following the European and International Directives for Clinical Research in order to strengthen the capacity of the European Union to study the determinants of ophthalmic diseases and to develop and optimise the use of diagnostic, prevention and treatment strategies in ophthalmology.

EVICR.net Eye Platform is a long-term initiative to establish a platform to gather high quality ophthalmology data generated in Europe and allow the secondary use of data in performing large data analysis and foster clinical research.

With this Eye Platform EVICR.net aims to provide technological solutions that allow overcoming privacy and regulation issues associated with the sharing of data from different institutions/countries, in a secure, easy to use manner.

With EVICR.net Eye Platform, the Members Sites will have the opportunity to participate in clinical research with secondary use data analysis; Authorship of publications and presentations of Results; the opportunity to propose new analysis to answer key research questions; and increase overall visibility and stature as researchers

Background:

On colour fundus photographs, drusen size and changes in retinal pigment epithelium are used to classify the severity of AMD into early, intermediate and advanced stages.Early AMD is characterised by medium sized drusen of 63 µm to 124 µm with no RPE changes. Intermediate AMD include large drusen (≥125 µm) or medium-sized drusen with pigmentary changes. These eyes with intermediate AMD have a high risk of progression to advanced AMD, including either geographic atrophy or exudative AMD due to macular neovascularisation (MNV). Visual deterioration is seen in these two advanced stages. Therefore, there is an unmet need to identify those at risk of disease progression to advanced AMD so that preventive options can be evaluated and implemented. However, a significant amount of research is required to better understand the risk of disease progression.

With the advent of multimodal imaging, there is growing evidence of new imaging markers of disease progression in eyes with intermediate AMD. For example, on infrared reflectance (IR), optical coherence tomography (OCT) and autofluorescence (AF), subretinal drusenoid deposits (SDD) are seen in some eyes with intermediate AMD and these have been identified as a predictor of fast progression to advanced AMD. Multimodal images have also shown that early atrophic changes may occur in intermediate AMD before the classical diagnosis of atrophy seen as hypoautofluorescence on AF. The Classification of Atrophy Meetings (CAM) group defined a few imaging characteristics as precursors of geographic atrophy and designated them together as incomplete retinal pigment epithelium and outer retinal atrophy (iRORA). A region of signal hypertransmission into the choroid of <250um, a corresponding zone of attenuation or disruption of the RPE, with or without the persistence of basal laminar deposits (BLamD) and evidence of overlying photoreceptor degeneration, i.e., subsidence of the inner nuclear layer (INL) and outer plexiform (OPL), presence of a hyporeflective wedge in the Henle fiber layer (HFL), thinning of the outer nuclear layer (ONL), disruption of the external limiting membrane (ELM), or disintegrity of the ellipsoid zone (EZ), and when these criteria do not meet the definition of complete retinal pigment epithelium and outer retinal atrophy (cRORA) that defines geographic atrophy on colour photographs. cRORA is defined as zone of hyper transmission of ≥250 µm, zone of attenuation or disruption of RPE band of ≥250 µm with evidence of overlying photoreceptor degeneration characterised by features that include outer nuclear layer (ONL) thinning, external limiting membrane (ELM) loss, and ellipsoid zone (EZ) or interdigitating zone (IZ) loss. Multimodal imaging also showed that drusen sizes on OCT are indeed larger than visualised on colour photographs. On en-face OCT, large drusen is defined as drusen diameter ≥145 µm, medium drusen diameters 100 µm to 144 µm, and small drusen diameters <100 µm. So, these markers and other novel imaging characteristics may better predict disease progression from intermediate AMD.However, a large multimodal image resource is required to develop such prediction models.

The Heidelberg Spectralis device enables multimodal imaging, and the OCT scans can be segmented by in-built automated Heidelberg software and manually corrected where necessary. So, a large database of Heidelberg imaging data of intermediate AMD will facilitate researchers to study the disease progression in detail.

ELIGIBILITY:
Inclusion Criteria:

Each dataset per patient should have one eye as the study eye with:

* Intermediate AMD with no atrophy and no subretinal drusenoid deposits
* Intermediate AMD with no atrophy with subretinal drusenoid deposits
* Intermediate AMD with early atrophy (iRORA) with no Subretinal drusenoid deposits
* Intermediate AMD with early atrophy (iRORA) with Subretinal drusenoid deposits
* Intermediate AMD with evidence of cRORA

Non-study eye images will not be exported but information about the status of the macula should be added using the following options:

* Established Geographic Atrophy (cRORA)
* Exudative AMD (presence of MNV)
* Early AMD
* Healthy macula

Exclusion Criteria:

* Both eyes have exudative AMD or geographic atrophy at baseline.
* Co-existent ocular disease: Any other ocular condition that, in the investigator's opinion, might affect or alter visual acuity during the study.
* Any patient who has opted out of their information being used for research nationally or locally at any Member Site.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with Age-related macular degeneration (AMD)
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of conversion to atrophy at two years | 24 months
  Number of patients who developed new or increasing atrophy

CONTACTS AND LOCATIONS:
Locations (25):
- Department of Ophthalmology, University Hospital, Nantes, Nantes, France
- Germany (6):
  - Department of Ophthalmology University of Bonn, Bonn
  - Department of Ophthalmology University of Freiburg, Freiburg im Breisgau
  - Department of Ophthalmology Justus/Liebig/University/Giessen, Giesen
  - Department of Ophthalmology St. Franziskus/Hospital Münster, Münster
  - Department of Ophthalmology University of Muenster Medical Center, Münster
  - Eye Clinic Sulzbach, Knappschaft Hospital Saar, Sulzbach
- Royal Victoria Eye and Ear Research Foundation, Dublin, Ireland
- Italy (3):
  - Medical Retina Service, Operative Unit Ophthalmology / MultiMedica Spa (IRCCSMM), Milan
  - Eye Unit, University Hospital Maggiore della Carità, Novara
  - Department of Ophthalmology University of Udine, Udine
- Department of Ophthalmology Radboud University Medical Centre Nijmegen, Nijmegen, Netherlands
- Portugal (4):
  - AIBILI-CEC (AIBILI- Clinical Trials Centre), Coimbra
  - Espaço Médico de Coimbra, Coimbra
  - Instituto de Oftalmologia Dr. Gama Pinto, Lisbon
  - Department of Ophthalmology Porto Medical School / Hospital S. João, Porto
- Spain (4):
  - Institut Català de Retina (ICR), Clinical Trial Unit, Barcelona
  - Institut de la Màcula Centro Médico Teknon, Barcelona
  - Valles Ophthalmology Research, S.L., Barcelona
  - Clínica Oftalmológica AIKEN / Fundación Aiken de la Comunitat Valenciana, Valencia
- Switzerland (2):
  - University Hospital Basel, University Eye Clinic, Basel, Basel
  - Swiss Visio Retina Research Center, Swiss Visio Montchoisi, Lausanne
- United Kingdom (3):
  - Clinical Trial Unit, Dep. Ophth., Gloucestershire Hospitals NHS Foundation Trust, Cheltenham
  - Clinical Eye Research Centre - St. Paul's Eye Unit, Royal Liverpool University Hospital, Liverpool
  - NIHR Moorfields Clinical Research Facility, Moorfields Eye Hospital, NHS Foundation Trust, London

REFERENCES:
- [Background] Ferris FL 3rd, Wilkinson CP, Bird A, Chakravarthy U, Chew E, Csaky K, Sadda SR; Beckman Initiative for Macular Research Classification Committee. Clinical classification of age-related macular degeneration. Ophthalmology. 2013 Apr;120(4):844-51. doi: 10.1016/j.ophtha.2012.10.036. Epub 2013 Jan 16. PMID 23332590
- [Background] Spaide RF, Ooto S, Curcio CA. Subretinal drusenoid deposits AKA pseudodrusen. Surv Ophthalmol. 2018 Nov-Dec;63(6):782-815. doi: 10.1016/j.survophthal.2018.05.005. Epub 2018 May 31. PMID 29859199
- [Background] Kim DY, Loo J, Farsiu S, Jaffe GJ. COMPARISON OF SINGLE DRUSEN SIZE ON COLOR FUNDUS PHOTOGRAPHY AND SPECTRAL-DOMAIN OPTICAL COHERENCE TOMOGRAPHY. Retina. 2021 Aug 1;41(8):1715-1722. doi: 10.1097/IAE.0000000000003099. PMID 33411474
- [Background] Sadda SR, Guymer R, Holz FG, Schmitz-Valckenberg S, Curcio CA, Bird AC, Blodi BA, Bottoni F, Chakravarthy U, Chew EY, Csaky K, Danis RP, Fleckenstein M, Freund KB, Grunwald J, Hoyng CB, Jaffe GJ, Liakopoulos S, Mones JM, Pauleikhoff D, Rosenfeld PJ, Sarraf D, Spaide RF, Tadayoni R, Tufail A, Wolf S, Staurenghi G. Consensus Definition for Atrophy Associated with Age-Related Macular Degeneration on OCT: Classification of Atrophy Report 3. Ophthalmology. 2018 Apr;125(4):537-548. doi: 10.1016/j.ophtha.2017.09.028. Epub 2017 Nov 2. PMID 29103793